CLINICAL TRIAL: NCT00195000
Title: Phase II Evaluation of Gemtuzumab Ozogamicin in Combination With Cytarabine in Untreated Patients Above the Age of 60 Years With Acute Myeloid Leukemia and High-Risk Myelodysplastic Syndrome
Brief Title: Mylotarg and Ara-C in Untreated Patients Above 60 Years With AML and High-Risk MDS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Eric Feldman, M.D., Weill Cornell Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0403-762
Record Dates: First submitted 2005-09-13; First posted 2005-09-19 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Acute Myeloid Leukemia; Myelodysplastic Syndrome
Keywords: Acute Myeloid Leukemia; Myelodysplastic Syndrome
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Gemtuzumab; Cytarabine

INTERVENTIONS:
Drug: Mylotarg — 6 mg/m2 on day 1
  Other Names: Gemtuzumab Ozogamicin
Drug: Cytarabine — 100 mg/m2 given as continuous infusion daily for 7 days.
  Other Names: Ara-C

SUMMARY:
The purpose of this study is to find out how safe and effective the combination of Mylotarg in combination with cytarabine is in treating patients with Acute Myeloid Leukemia and advanced Myelodysplastic Syndrome over the age of 60 years.

DETAILED DESCRIPTION:
To evaluate the safety and efficacy of gemtuzumab ozogamicin in combination with cytarabine in inducing complete remission in patients with AML and advanced MDS over the age of 60 years.

Patients eligible for treatment will receive the following:

Mylotarg at 6 mg/m2 on day 1 as a 2 hour intravenous infusion

Cytarabine at 100 mg/m2/day as a continuous intravenous infusion daily for 7 days

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of AML or advanced MDS
* No prior cytotoxic treatment for AML. (patients may have been treated with prior biologic therapy) Patients with MDS or AML that has evolved from MDS, could have received prior low-dose cytotoxic therapy (i.e. azacytidine or low-dose ara-C).

Exclusion Criteria:

* Uncontrolled or severe cardiovascular disease or pulmonary disease

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2003-05; Primary Completion 2006-05 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and efficacy of gemtuzumab ozogamicin (Mylotarg) in combination with cytarabine in inducing complete remission in patients with AML and advanced MDS over the age of 60 years. | From entry until 30 days post treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Feldman, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medcial College of Cornell University, New York, New York, United States